CLINICAL TRIAL: NCT06783803
Title: Application of Linkage Analysis in the Identification of Novel Hereditary Factors in Familial Aneurysms
Acronym: ORPHADIAG
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Alessandro Pini, Pincipal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: ORPHADIAG
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Familial Thoracic Aortic Aneurysm and Aortic Dissection
Keywords: familial thoracic aortic aneurysm and dissection; Linkage analysis; biomarkers
MeSH Terms: conditions — Aortic Aneurysm, Familial Thoracic 1 | interventions — Genetic Linkage

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Whole Exome Sequencing (WES) of peripheral blood of patients with FTAAD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- FTAAD: members of families with FTAAD
  Interventions: Diagnostic Test: Linkage Analysis

INTERVENTIONS:
Diagnostic Test: Linkage Analysis — WES-Linkage analysis in families with FTAAD in follow-up in an Italian reference centre for genetic aorthopathies

SUMMARY:
The aim of this study is to describe the effectiveness of the application of Linkage Analysis, compared to the standard procedures currently provided by the italian NHS, in the identification of thoracic aortic aneurysms and dissection (TAAD) transmission markers in individuals with familial TAAD.

DETAILED DESCRIPTION:
According to current guidelines, it is important to screen first-degree relatives of patients with familial thoracic aortic aneurysm and dissection (FTAAD) using imaging techniques in order to detect any undiagnosed or asymptomatic cases. The current diagnostic methods for FTAAD involve clinical and instrumental diagnosis. In addition to these methods, genetic analysis through DNA testing, using a blood sample has become an essential tool. The use of massive parallel sequencing (NGS) of multiple genes or the entire exome (Whole Exome Sequencing - WES) is considered the gold standard for genetic diagnosis of FTAAD. However, it should be noted that linkage studies are not currently included in the diagnostic protocols of the Italian National Health System, although they may be helpful in complex familial cases where DNA sequencing has not provided conclusive evidence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ascending thoracic aortic aneurysms in the absence of a mutation identified by WES
* Subjects with small and medium artery aneurysms in the absence of a mutation identified by WES
* Relatives of individuals with ascending thoracic aortic aneurysms in the absence of a mutation identified by WES
* Relatives of individuals with ascending thoracic aortic aneurysms in the absence of a mutation identified by WES
* Signed informed consent

Exclusion Criteria:

* Subjects wit syndromic FTAAD with WES identified gene mutation
* Subjects wit non-syndromic FTAAD with WES identified gene mutation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Families of patients with FTAAD in follow-up in an italian reference centre for genetic aorthopathies.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
DNA sequences in FTAAD | 16 months
  Identify those chromosome regions containing the DNA sequences responsible for each enrolled member of FTAAD families

SECONDARY OUTCOMES:
Mutations associated with Mendelian and monogenic diseases | 24 months
  Identification of potential sites for the location of the responsible gene and mutations associated with Mendelian and monogenic diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Genetic Centre, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
IPD will be considered for sharing after data collection and analysis

REFERENCES:
- [Background] Isselbacher EM, Lino Cardenas CL, Lindsay ME. Hereditary Influence in Thoracic Aortic Aneurysm and Dissection. Circulation. 2016 Jun 14;133(24):2516-28. doi: 10.1161/CIRCULATIONAHA.116.009762. PMID 27297344
- [Background] Carino D, Agostinelli A, Molardi A, Benassi F, Gherli T, Nicolini F. The role of genetic testing in the prevention of acute aortic dissection. Eur J Prev Cardiol. 2018 Jun;25(1_suppl):15-23. doi: 10.1177/2047487318756433. PMID 29708033